CLINICAL TRIAL: NCT06409728
Title: Prevalence and Healthcare Consumption of ASD Patients Using French Medico-administrative Data (SNDS)
Brief Title: Prevalence and Healthcare Consumption of ASD Patients Using French Medico-administrative Data
Acronym: ECO-TSA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0063
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Administrative claims; Population surveillance
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Autism Spectrum Disorder (ASD) is one of the neurodevelopmental disorders described in the DSM5 (American Psychiatric Association, 2013). This heterogeneous syndrome appears in childhood and persists throughout life with different developments from one individual to another. It is clinically characterized by the combination of deficits in social communication with restricted and repetitive behaviors. The prevalence of ASD has seen a significant increase over the last 10 years, with estimates varying greatly from one country to another, ranging from 4.2/1,000 in France to 31/1,000 in Iceland. In France, prevalence has been estimated by two child disability registers set up in the departments of Haute-Garonne (RHE31), Isère, Savoie, and Haute-Savoie (RHEOP), but there is no epidemiological surveillance system to estimate the national prevalence of ASD in the general population. However, the production of reliable epidemiological data at the national and territorial levels is essential for addressing the needs of individuals with ASD and for evaluating public policies.

The main objective of our project is to estimate the annual prevalence of ASD in children, adolescents, and young adults at the national and regional levels using medico-administrative databases (SNDS), to study its evolution over the period 2010-2019 and its geographical distribution in relation to socio-demographic indicators and healthcare accessibility. Our secondary objectives are to validate an algorithm for detecting ASD in the National Health Data System (SNDS) and to estimate the direct medical costs associated with ASD management.

The SNDS databases contain all medical care and treatments reimbursed for Health Insurance beneficiaries provided in the private or public sector. A case detection algorithm will be tested and validated on validation samples. Then, the prevalence of ASD will be estimated, taking into account geographical, socio-economic, and healthcare accessibility indicators, in order to study the factors associated with the significant disparity in rates observed in France and abroad. An estimate of direct medical costs will be made from the health insurance perspective.

Our project therefore proposes the development of reliable indicators on the management of ASD in France with the aim of providing useful indicators and tools for guiding health and disability policies in France, promoting the development of appropriate interventions, and thus contributing to the improvement of the care and support of individuals with ASD as well as reducing inequalities in access to healthcare for these vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 16 years or younger
* For case : with an ICD-10 code for ASD (F84*)
* For control : without an ICD-10 code for ASD (F84*)

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Population Study are children aged 16 or younger with ASD hospitalized in unversity hospital.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
ASD diagnostic code in healthcare database | 1 year
  ≥ 1 hospitalization with ASD diagnostic code (F84*)

SECONDARY OUTCOMES:
Prevalence of ASD | 2010-2019
Cost of medical care reimbursed by health insurance for patient with ASD | 2010-2019

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University Hospital Dijon, Dijon
  - University Hospital Montpellier, Montpellier